CLINICAL TRIAL: NCT01676740
Title: Randomized Ttrial to Establish the Efficacy of Hematinic Agents in Patietns With Mild Anemia Undergoing Total Hip or Knee Replacement in Avoiding Blood Transfusion
Brief Title: Iron and Vitamin Adminstration Prior to Joint Replacement to Prevent Transfusion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, Martin Ellis, Head Hematology Institute, Meir Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MMCHI0112
Record Dates: First submitted 2012-08-29; First posted 2012-08-31 (Estimated); Last update posted 2012-09-03 (Estimated); Status verified 2012-08

CONDITIONS: Excessive Amount of Blood / Fluid Transfusion
Keywords: hematinic therapy; blood transfusion; joint replacement
MeSH Terms: interventions — Iron-Dextran Complex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Mild anemia, normal hematinics (Placebo Comparator): Mild anemia, normal iron studies, serum folate and vitamin B12 levels - will receive placebo
  Interventions: Drug: Placebo
- Anemia, normal hematinics (Experimental): Mild anemia, deficient iron, folate or vitamin B12 levels Iron supplement will be given
  Interventions: Drug: Iron Supplement,
- Deficeicnt hematinics (Other): Iron supplement will be provided
  Interventions: Drug: Iron Supplement,

INTERVENTIONS:
Drug: Iron Supplement, — Pills to be swallowed
  Other Names: Ferrifol
  Arms: Anemia, normal hematinics; Deficeicnt hematinics
Drug: Placebo — Daily administration of active drug or placebo
  Arms: Mild anemia, normal hematinics

SUMMARY:
To establish the efficacy of screening for anemia and treatment of mild anemia with iron and vitamins prior to THR and TKR as a means of increasing hemoglobin and reducing perioperative allogeneic blood transfusion.

DETAILED DESCRIPTION:
Patients with mild anemia will be identified at preoperative clinic visit

* Patients will be screened for inclusion and exclusion criteria
* Eligible patients will have laboratory testing performed as follows: CBC, liver and kidney function tests, serum iron, transferrin, ferritin, serum folic acid, vitamin B12 and C-reactive protein
* Patients will be assigned to a deficient group or non-deficient group depending upon laboratory hematinic values
* Patients in the "non-deficient' group will be randomized using a computer-generated code to treatment or no treatment
* Treatment will begin within 2 weeks of laboratory testing and 4-6 weeks prior to surgery.
* Hematinic therapy will consist of oral ferric hydrochloride polymaltose 200 mg/d and folic acid 0.4 mg/d; sublingual vitamin B12 1000 µg three times a week
* On the day of surgery laboratory testing will be performed as follows: CBC, kidney and liver function tests, serum iron, transferrin, ferritin, serum folic acid, vitamin B12 and C-reactive protein.
* The same surgical team in each center will operate on all study patients and will be blinded to the preoperative hemoglobin
* Routine postoperative management will be provided as determined by the treating physicians
* Blood transfusion will be decided upon by a study physician at each center blinded to the patients' group assignment and preoperative hemoglobin
* The primary outcome will be perioperative blood transfusion (from 24 hours prior to surgery until hospital discharge)
* Secondary outcomes will be length of hospitalization, postoperative wound infection, walking ability across room at 30 days

ELIGIBILITY:
Inclusion Criteria:

* Age > 50 years
* Ability to provide informed consent
* Elective THR or TKR
* Mild anemia: Hematocrit 29-39% in men, 29-36% in women

Exclusion Criteria:

* Identified cause of anemia excluding hematinic deficiency
* Known source of blood loss
* Known coagulopathy
* Unstable coronary syndrome in the previous 3 months
* Pathologic fracture, presence of malignancy
* Repeat THR or TKR
* Orthopedic trauma within the previous 3 months
* ASA class ≥ 4
* Creatinine clearance < 30 ml/min
* AST/ALT > 2x upper limit of normal
* Preexisting use of hematinic agents
* Planned acute normovolemic hemodilution
* Refusal to receive blood products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2012-11; Primary Completion 2013-12 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
Perioperative blood transfusion | 1 day prior to surgery until hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Martin H Ellis, MD, Principal Investigator — Meir Medical Center
Locations (1):
- Meir Medical Center, Kfar Saba, Israel